CLINICAL TRIAL: NCT03062644
Title: A Randomized, Double-Blind, Multicenter, Placebo- and Active Comparator-Controlled Study to Evaluate Efficacy and Safety of MR308 in the Treatment of Acute Pain After Abdominal Hysterectomy Surgery Under General Anaesthesia (STARDOM2).
Brief Title: Efficacy and Safety in a Randomised Acute Pain Study of MR308: STARDOM2.
Acronym: STARDOM2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MR308-3502
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Acute Pain
Keywords: Open Total or Subtotal Abdominal Hysterectomy
MeSH Terms: conditions — Acute Pain | interventions — Tramadol; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MR308 100 mg bid (Experimental): Tramadol/Celecoxib)
  Interventions: Drug: MR308
- MR308 150 mg bid (Experimental): Tramadol/Celecoxib
  Interventions: Drug: MR308
- MR308 200 mg bid (Experimental): Tramadol/Celecoxib
  Interventions: Drug: MR308
- Tramadol 100 mg qid (Active Comparator): Tramadol
  Interventions: Drug: MR308
- Celecoxib 100 mg bid (Active Comparator): Celecoxib
  Interventions: Drug: MR308
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: MR308

INTERVENTIONS:
Drug: MR308 — two times daily; Mode of Administration:oral
  Other Names: Tramadol/Celecoxib
  Arms: MR308 100 mg bid; MR308 150 mg bid; MR308 200 mg bid
Drug: MR308 — four times daily; Mode of Administration:oral
  Other Names: Tramadol
  Arms: Tramadol 100 mg qid
Drug: MR308 — two times daily; Mode of Administration:oral
  Other Names: Celecoxib
  Arms: Celecoxib 100 mg bid
Drug: MR308 — given four times daily to maintain the blind; Mode of Administration:oral
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
The MR308-3502 study is a multicenter double-blind, randomised, placebo- and active comparator-controlled study in female subjects to evaluate the efficacy and safety of MR308 with acute pain after TAH or STAH (total or subtotal abdominal hysterectomy).

DETAILED DESCRIPTION:
This is a multicenter double-blind, randomised, placebo- and active comparator-controlled study in female subjects to evaluate the efficacy and safety of MR308 with acute pain after total or subtotal abdominal hysterectomy (TAH or STAH).

The screening Visit (Visit 1) can take place up to 28 days before the planned TAH or STAH. The surgery will be performed at Visit 2. Visit 2 consists of three different sections, a part before the surgery, the surgery and post surgery. On the next Day (Visit 3) subjects will qualify for further participation by regular measurements of their pain. Subjects meeting all eligibility criteria, such as defined pain levels, will be randomised to one of six treatment groups and be given IMPs for 120h. Subjects who will not be randomised are screen failures and will be given standard care as per local practice.

Visits 4, 5, 6 ,7 and 8, one to five days after randomisation will be performed to record efficacy and safety parameters.

The last dose of IMP should be taken by the subject about 120h after the initial dose and before Visit 8 (Completion/Discontinuation Visit) is performed.

The Adverse Event (AE) Follow up Visit (Visit 9) is the last study visit and should not be done earlier than seven days after the subject's last dose of IMP. It can be performed by telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ≥ 18 years on the day of consent.
2. Willing and able to provide written informed consent for this study.
3. Subjects are scheduled to have a total or subtotal abdominal hysterectomy under general anasethesia via a Pfannenstiel incision.
4. The elective procedure (total or subtotal hysterectomy with or without salpingo-oophorectomy) must be for benign conditions within 28 days of screening. Subjects with stage 0 carcinoma in situ of cervix, endometrial hyperplasia or clinically staged 1A or 1B endometrial cancer are allowed to participate.
5. American Society Anaesthesiology physical status of I or II.
6. If a female is of child-bearing potential, she must be using highly effective methods of contraception throughout the study, not breastfeeding, and have negative pregnancy tests prior to receiving IMP. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner).
7. Good general health as judged by Investigators on the basis of medical history and physical examination.
8. Willingness to comply with the study procedures and requirements.

Additional Inclusion Criteria after Surgery:

1. Abdominal hysterectomy completed without any immediate complication.
2. Tolerating oral fluids, no uncontrolled nausea/vomiting and ready to take oral analgesia.
3. The subject is alert and calm, spontaneously pays attention to caregiver, e.g. RASS = 0 (Sessler et al., 2002 & Ely et al., 2003).
4. Subjects will be capable to sit up from supine, stand up from a sitting position and walk 10 meters without assistance in the morning of the day following surgery.
5. Subjects with moderate or severe pain (qualifying PI-VAS score ≥ 45mm and < 70mm or ≥ 70mm and ≤ 90mm) as a result of a surgical procedure (abdominal hysterectomy) under general anaesthesia. This must be measured within a maximum of 24 hours after leaving the recovery room and subjects can only be randomised on the day after surgery, after cessation of the post-operative analgesia.

Exclusion Criteria:

1. Any abnormal laboratory value that is clinically significant in the opinion of Investigator that would compromise the safety of the subject in the study.
2. Any recent history of frequent nausea or vomiting, dizziness within the last 3 months regardless of etiology.
3. Subjects having any medical condition or treatment that is either a warning or contraindication as per the SmPC of tramadol (e.g. selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, MAO inhibitors (within 14 days before taking IMP), antipsychotics, anticonvulsant and other seizure threshold-lowering medicinal products), celecoxib (e.g. increased risk of post-operative bleeding, active peptic ulceration, GI bleeding or inflammatory bowel disease) or paracetamol.
4. Known sensitivity and/or contraindication to tramadol, celecoxib, paracetamol, sulfonamides, opioids, NSAIDS, COX-2 inhibitors, or related compounds or formulation excipients as well as severe hypersensitivity reactions (e.g. anaphylactic shock, bronchospasm, angioedema) to any drugs.
5. Subjects who are known to have had inadequate pain relief from paracetamol, tramadol or celecoxib.
6. Subjects requiring any medication which is prohibited as per section prohibited medication.
7. Subjects who are in the Investigator's opinion considered at increased risk of operative (those associated with the surgical procedure and general anaesthesia) and post-operative complications, e.g. excessive post-operative bleeding, infection.
8. Any history of drug or alcohol abuse, misuse, physical or psychological dependence, mood changes, sleep disturbance and functional capacity which have an impact on pain perception.
9. Significant neurological or psychiatric disorders including mental instability (unrelated to the pain) that could interfere with pain assessment; other pre-existing or new non-abdominal/pelvic pain that might impair the assessment of the nociceptive pain.
10. Any medical history of significant and/or inadequately controlled cardiovascular (uncontrolled high blood pressure, high risk of cardiovascular events, severe heart failure), pulmonary, hematologic, (including coagulopathy/bleeding disorders), neurological (e.g. subjects with epilepsy or those susceptible to seizures), liver disease (e.g. severe hepatic impairment), kidney disease (e.g. serum creatinine level greater than 1.5 times the upper limit of normal, impaired renal function in subjects taking diuretics, ACE-inhibitors, or angiotensin II antagonists), endocrine, immunologic, dermatologic painful conditions or any other conditions that may compromise the ability of the subject to participate in the study or might interfere with drug absorption, distribution, metabolism or excretion.
11. Previous randomisation in this study.
12. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period).
13. Subjects who were treated regularly with opioid analgesic or NSAIDs within 30 days prior to screening or who have received a long-acting NSAID within three days prior to the start of the surgery.
14. Subjects who are incapable of complying with the protocol.
15. Epidural or spinal anaesthesia or infiltration of the wound with an infusion of a local anaesthetic agent is not allowed. A single perioperative dose is allowed.
16. History or ongoing chronic pelvic inflammatory disease or painful endometriosis.
17. History of advanced gynaecological cancers.

Additional Exclusion Criteria after Surgery:

1. Serious complication during surgery and up to randomisation, including:

   * Post-operative primary and secondary bleed that cannot be controlled.
   * Subjects who have not had the abdominal hysterectomy surgery completed as planned.
2. If in the Investigator's opinion, there are any factors that may affect compliance with the protocol.
3. Subject clinical need for antiemetics (apart from standard perioperative practice as defined in the protocol) or any other medication which is prohibited as per section prohibited medication.
4. Subjects who have received any analgesic medication other than perioperative analgesia as described in the protocol.
5. Any concerns that renal function has deteriorated, e.g. a laboratory parameter, profound hypotension, poor urine output or excessive bleeding during surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1138 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of MR308 doses in the treatment of moderate to severe acute pain, based on the Sum of Pain Intensity Differences (SPID) from 0-4 hours. | 0-4 hours
  The primary efficacy endpoint is the Sum of Pain Intensity Differences over 0-4 hours (SPID4). SPID4 is derived as the weighted Sum of Pain Intensity Differences (baseline pain - current pain), measured at different time points via the PI-VAS. Time between two consecutive measurements will be used for weighting. Larger values indicate larger pain relief.

CONTACTS AND LOCATIONS:
Locations (8):
- Minsk City Gynecology Hospital Department of Gynecology, Minsk, Belarus
- "Multiprofile Hospital for Active Treatment - Doverie" AD, Sofia Department of Gynecology, Sofia, Bulgaria
- Victoria Hospital - London Health Sciences Centre, London, Ontario, Canada
- Bajcsy-Zsilinszky Korhaz Szuleszet-Nogyogyaszati Osztaly, Budapest, Hungary
- Vidzeme Hospital Department of Gynecology and Obstetrics, Valmiera, Latvia
- Wojewódzki Szpital im. Św. Ojca Pio w Przemyślu Oddział Ginekologii i Położnictwa, Przemyśl, Poland
- Federal State Budgetary Institution National Medical-Surgical Centre named after N.I. Pirogov of the Ministry of Health of the Russian Federation Anesthesiology, Moscow, Russia
- Hospital Universitari Germans Trias i Pujol Anestesia y Reanimación, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viscusi ER, Langford R, Morte A, Vaque A, Cebrecos J, Sust M, Gimenez-Arnau JM, de Leon-Casasola O. Safety of Co-Crystal of Tramadol-Celecoxib (CTC) in Patients with Acute Moderate-to-Severe Pain: Pooled Analysis of Three Phase 3 Randomized Trials. Pain Ther. 2024 Dec;13(6):1617-1631. doi: 10.1007/s40122-024-00655-w. Epub 2024 Sep 24. PMID 39316284
- [Derived] Langford R, Morte A, Sust M, Cebrecos J, Vaque A, Ortiz E, Fettiplace J, Adeyemi S, Raba G, But-Husaim L, Gascon N, Plata-Salaman C. Efficacy and safety of co-crystal of tramadol-celecoxib (CTC) in acute moderate-to-severe pain after abdominal hysterectomy: A randomized, double-blind, phase 3 trial (STARDOM2). Eur J Pain. 2022 Nov;26(10):2083-2096. doi: 10.1002/ejp.2021. Epub 2022 Sep 24. PMID 35974668